CLINICAL TRIAL: NCT06289764
Title: The Effect of Aromatherapy Application With Bergamot and Grapefruit Essential Oils on Premenstrual Syndrome and Menstrual Symptoms
Brief Title: The Effect of Aromatherapy Application With Bergamot and Grapefruit Essential Oils on PMS
Acronym: Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra ÖZER (Other)
Collaborators: KTO Karatay University (Other)
Responsible Party: Sponsor-Investigator, Esra ÖZER, Assist Prof, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 7/02/2024/131
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Premenstrual Syndrome-PMS
Keywords: Aromatherapy; Premenstrual syndrome; Menstrual symptom
MeSH Terms: conditions — Premenstrual Syndrome | interventions — almond oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sweet almond oil (Placebo Comparator): Premenstrual symptom scale will be applied to the participants who volunteered to participate in the study. Aromatherapy will be applied to people with a premenstrual symptom score exceeding 110. 3 groups will be formed from people with pms symptoms. 1st group will receive Bergamot essential oil, 2nd group will receive Grapefruit essential oil, 3rd group (placebo group) will receive sweet almond oil. Selected women will be allowed to smell 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. The aromatic oil will be put 3 drops on a cotton ball and the participants will smell it. Participants will be allowed to inhale the scent for 30 minutes in the fowler position at a distance of 15 cm.
  Interventions: Other: Sweet almond oil
- Bergamot essential oil (Experimental): Premenstrual symptom scale will be applied to the participants who volunteered to participate in the study. Aromatherapy will be applied to people with a premenstrual symptom score exceeding 110. 3 groups will be formed from people with pms symptoms. 1st group will receive Bergamot essential oil, 2nd group will receive Grapefruit essential oil, 3rd group (placebo group) will receive sweet almond oil. Selected women will be allowed to smell 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. The aromatic oil will be put 3 drops on a cotton ball and the participants will smell it. Participants will be allowed to inhale the scent for 30 minutes in the fowler position at a distance of 15 cm
  Interventions: Other: Bergamot Essential Oil
- Grapefruit essential oil (Experimental): Premenstrual symptom scale will be applied to the participants who volunteered to participate in the study. Aromatherapy will be applied to people with a premenstrual symptom score exceeding 110. 3 groups will be formed from people with pms symptoms. 1st group will receive Bergamot essential oil, 2nd group will receive Grapefruit essential oil, 3rd group (placebo group) will receive sweet almond oil. Selected women will be allowed to smell 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. The aromatic oil will be put 3 drops on a cotton ball and the participants will smell it. Participants will be allowed to inhale the scent for 30 minutes in the fowler position at a distance of 15 cm
  Interventions: Other: Grapefruit Essential Oil

INTERVENTIONS:
Other: Bergamot Essential Oil — Selected women will be smelled 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. Application will be repeated for 3 cycles.
  Arms: Bergamot essential oil
Other: Grapefruit Essential Oil — Selected women will be smelled 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. Application will be repeated for 3 cycles.
  Arms: Grapefruit essential oil
Other: Sweet almond oil — Selected women will be smelled 3 times a day, at the same time every day, for 4 days, within 7 days before menstruation. Application will be repeated for 3 cycles
  Arms: Sweet almond oil

SUMMARY:
Aromatherapy is;the science of using highly concentrated essential oils or essences distilled from plants to take advantage of their therapeutic properties. Essential oils or essences are obtained from various parts of plants (root, leaf, flower, bark, fruit) and used therapeutically for physical and psychological well-being.

Premenstrual syndrome (PMS) is a health problem characterized by the periodic occurrence of physical, cognitive, emotional and behavioral symptoms during the luteal phase of the menstrual cycle, ending with the onset of menstruation or with the alleviation of symptoms within a few days after the onset of menstruation. It is reported that approximately 80-95% of women complain of PMS complaints.

Although the use of aromatherapy in womens health is widespread, there is no study comparing bergamot and grapefruit essential oils. The aim of this study was to determine the effect of aromatherapy with bergamot and grapefruit essential oils on premenstrual syndrome and menstrual symptoms.

DETAILED DESCRIPTION:
Aromatherapy is the science of using highly concentrated essential oils or essences distilled from plants to take advantage of their therapeutic properties. Essential oils or essences are obtained from various parts of plants (root, leaf, flower, bark, fruit) and used therapeutically for physical and psychological well-being.The fact that aromatherapy is a noninvasive procedure and is easy to use allows aromatherapy to be widely used . Aromatic oils can be applied in four basic ways. These are topical (touch, compress or bath), internal (mouthwash, vaginal or anal suppositories), oral (capsules or dilution in honey, alcohol or diluent) and inhalation (direct or indirect inhalation with or without steam). Essential oils, which can be applied in various ways, can directly reach the neocortex part of the brain through connections from the limbic system to the hypothalamus via odor. As a result of the effect of aromatic oils on the central nervous system, relaxation, sedation or stimulating effects occur, and thanks to the information flow reaching the brain with the stimulation of the central nervous system, the energy blockage in the body is broken and energy is released as a result. The healing process is supported by the balanced spread of the energy flow to the relevant organs, and physical and mental well-being emerges. Aromatherapy is used in many health fields as well as in womens health.

Premenstrual syndrome (PMS) is a health problem characterized by periodic physical, cognitive, emotional and behavioral symptoms that occur periodically during the luteal phase of the menstrual cycle, ending with the onset of menstruation or with the alleviation of symptoms within a few days after the onset of menstruation. It is stated that approximately 80-95% of women complain of PMS complaints. In studies in the literature, aromatherapy with various essential oils (rose, geranium, sage, lavender) was applied to women complaining of PMS complaints and it was determined that aromatherapy application had both psychological and physical positive effects by stating that depression, anxiety, anxiety, irritability, and pain perception decreased.

Menstrual symptoms are recognized as one of the biggest problems that negatively affect the health status and quality of life among women of reproductive age worldwide. Menstrual symptoms such as dysmenorrhea, heavy menstrual bleeding and mood disorders during the premenstrual period are known to be common in the general population. Menstrual symptoms affect womens activities of daily living and quality of life. In studies in the literature, aromatherapy with various essential oils (rose, sage, ginger) was applied to women with dysmenorrhea, but no study was found in which all menstrual symptoms were measured.

Bergamot (Citrus aurantium bergamia), a small tree belonging to the Rutaceae family among citrus fruits, grows in the Mediterranean region and is especially native to the southern coast of Italy. Bergamot essential oil (BEO) is an essential oil produced by extracting the fruit from the rind by cold pressing procedure or steam distillation. Bergamot essential oil has analgesic, sleep quality enhancing, relaxation, anti-inflammatory and antidepressant effects.

Grapefruit, one of the citrus families with the largest production in the world, is famous for its taste and nutritional value, and grapefruit essential oil has antibacterial, antimicrobial, antiseptic, antidepressant, anti-edema and appetite regulating effects.

Although the use of aromatherapy in womens health is widespread, no study comparing bergamot and grapefruit essential oil has been found. The aim of this study is to determine the effect of aromatherapy application with bergamot and grapefruit essential oils on premenstrual syndrome and menstrual symptoms.

ELIGIBILITY:
Inclusion Criteria

* To be between the ages of 18-35
* Experiencing at least 5 of the pms complaints (self-report)
* Not having respiratory diseases such as asthma and bronchitis (self-report)
* No pregnancy or suspected pregnancy (self-report)
* Not being allergic to any substance (self-report)
* Not having a systemic disease such as diabetes, hypertension (self-report)

Exclusion Criteria:

* Under 18, over 35 years of age Not experiencing pms complaints Finding anosmia Presence of respiratory system diseases Allergic symptoms to aromatherapy Being pregnantHaving a chronic disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Premenstrual syndrome scale (PMS) | Baseline and three months later
  It is a five-point Likert type scale consisting of 44 questions measuring the severity of premenstrual symptoms. A minimum of 44 and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates that the intensity of PMS symptoms increases. In the PMS scale, PMS is considered to be "present" if it exceeds 50% (110) of the total scale score (220).

SECONDARY OUTCOMES:
Menstrual Symptom Scale | Baseline and three months later
  Scale items are numbered according to the allocated factors for ease of use. 1-13. Items belong to the "Negative effects/somatic complaints" subscale, items 14-19. The items refer to the "Menstrual pain symptoms" subscale and items 20-22. The items belong to the "Coping methods" sub-dimension. Cronbach's Alpha value is 0.86. It is a five-point Likert type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. Average score for sub-dimensions Its increase indicates that the severity of menstrual symptoms related to that sub-dimension increases.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Ö ÖZER, Assist Prof., Principal Investigator — Ankara Medipol Unıversty
Locations (1):
- Ankara Medipol Unıversty, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be planned after the study is completed.

REFERENCES:
- [Derived] Ozer E, Doner SI, Dag Tuzmen H. The effect of aromatherapy intervention with Bergamot and Grapefruit essential oils on premenstrual syndrome and menstrual symptoms: a randomized controlled trial. BMC Complement Med Ther. 2025 May 1;25(1):162. doi: 10.1186/s12906-025-04857-3. PMID 40312670